CLINICAL TRIAL: NCT06268548
Title: Effect of Manual Diaphragmatic Activation on Diaphragm Function in Patients With Gastroesophageal Reflux Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shimaa Goda Sherif Ali, Demonstrator of physical therapy department for cardiothoracic/respiratory disorder & geriatric, faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004790
Record Dates: First submitted 2024-02-04; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-12

CONDITIONS: Diaphragm Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Experimental): Experimental , diaphragmatic activation with medical treatment ,15patients with gastroesophageal reflux disease do manual diaphragmatic activation in additional to traditional medical treatment
  Interventions: Other: Manual diaphragmatic activation
- Control (No Intervention): 30 patients with gastroesophageal reflux disease taking traditional medical treatment only

INTERVENTIONS:
Other: Manual diaphragmatic activation — Manual diaphragm release on diaphragm
  Arms: Study

SUMMARY:
This study was conducted to investigate Effect of manual diaphragmatic activation on diaphragm function in patients with gastroesophageal reflux disease

DETAILED DESCRIPTION:
Thirty both gender patients with gastroesophageal reflux disease enrolled in this study , study group And control group. To investigate Effect of manual diaphragmatic activation on diaphragm function in patients with gastroesophageal reflux disease

ELIGIBILITY:
Inclusion Criteria:

* patients with gastroesophageal reflux disease.
* the age will be ranged from 20 to 50 .
* body mass index from 20 to 34,9 kg/m2 .
* low level of physical therapy

Exclusion Criteria:

* Pregnancy
* open wound
* abdominal or spinal surgery
* Congenital or acquired disorder

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Both gender patients
Enrollment: 30 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-02-27 (Estimated)

PRIMARY OUTCOMES:
Diaphragm Excursion | 2 months
  Diaphragm Excursion

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No